CLINICAL TRIAL: NCT06706024
Title: Effect of a Breathing Exercise on Respiratory Function and 6-Minute Walking Distance in Patients Under Hemodialysis
Brief Title: Effect of a Breathing Exercise in Patients Under Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Seher Gönen Şentürk, PhD, RN, Assist. Prof., Çankırı Karatekin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 28-06-2022/26
Record Dates: First submitted 2024-03-18; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Breathing Exercise
Keywords: hemodialysis patient; breathing exercise program; nursing care
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study with a single group pretest-posttest design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- respiratory exercise program (Experimental): A practical explanation was given about how to use the flow-oriented Intensive Spirometry Device (ICC) (Triflow) after the 3rd hour of the treatment in the HD unit. Each of the patients was given the same brand and model flow-focused intensive spirometer (Triflow) device for breathing exercise.
  Interventions: Other: breathing exercise

INTERVENTIONS:
Other: breathing exercise — Patients Under Hemodialysis
  Other Names: 6 minute walking test

SUMMARY:
Purpose: To examine the effects of breathing exercises on respiratory functions and 6 Minute Walk Test (6 WT) distance in patients receiving hemodialysis treatment.

Method: This is a quasi-experimental study with a single group pretest-posttest design. It was conducted with 30 individuals in the hemodialysis unit of a public hospital between July 2022 and October 2022. Data were also collected before starting the intervention (week 1) and after completing the intervention (week 8). Socio-Demographic Data Survey, 6 Minute Walk Test and Respiratory Function Test were used as data collection tools and data were collected face to face. In the analysis of the data, mean, standard deviation, percentage, t test in dependent groups, and Wilcoxon analysis were used.

KeyWords: Individuals receiving hemodialysis treatment, respiratory exercise program, nursing care

DETAILED DESCRIPTION:
Creating and Implementing an Exercise Program Data were collected before starting the intervention (1st week) and after the intervention was completed (8th week). 6 Minute Walking Test and Respiratory Function Test were applied to the patients before the implementation of the exercise program and after 8 weeks of application. According to the results of the Pulmonary Function Test evaluated by the pulmonologist, COPD is in Grades 3 and 4. Stage 1 patients were not included in the study. A practical explanation was given about how to use the flow-oriented Intensive Spirometry Device (ICC) (Triflow) after the 3rd hour of the treatment in the HD unit. Each of the patients was given the same brand and model flow-focused intensive spirometer (Triflow) device for breathing exercise. The Triflow device has three compartments with a capacity of 1200 ml, with a ball of different colors in each compartment. The Triflow device is based on the patient taking a maximal inspiration, then holding the breath for as long as he can (at least 5 seconds), and then exhaling slowly. The patient watches the movement of the balls for visual feedback.

During Triflow use, patients were placed in a sitting position. They were told to hold the device in an upright position, put the mouthpiece of the Triflow in their mouth, completely cover the mouthpiece with their lips to prevent air from escaping, take a deep and slow breath after a quiet exhalation, increase the duration of holding their breath as much as the patient can tolerate, and then release the balls by exhaling. Patients were instructed to bring their devices with them to each session. Since some patients forgot their hemodialysis unit and exercise device and stated that they had difficulty in bringing them back and forth due to the long distance between the dialysis unit and home, each patient was given a special triflo device to be kept in the hemodialysis unit, separate from the ones they use at home.

The exercise program was performed 3 times a week for 8 weeks, under the supervision of the researcher, with 10 repetitions at the 3rd and 4th hours of the dialysis treatment. It was recommended that they do 10 repetitions every hour after waking up on days when there was no dialysis session. In the study, patients adhered to the breathing exercise program, and no problems were reported regarding device use during the session or at home.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥18 years old;
* Receiving HD treatment three times a week for at least 3 months;
* Not having a condition that prevents walking;

Exclusion Criteria:

* Having a history of Myocardial Infarction or Anginapectoris within the last month,
* Uncontrolled arrhythmia and heart rate >120/min,
* Having uncontrolled hypertension (BP>180/100 mm-Hg),
* Having a history of cerebrovascular accident
* Having advanced stage COPD (Stage 3, Stage 4) and advanced Stage Heart Failure (Stage 3/Stage 4),
* Having profound anemia (Hb<7 g/dl),
* Having a history of blood transfusion in the last month,
* Having an active and chronic infection (Tuberculosis, osteomyelitis, rheumatoid arthritis),
* Needing additional oxygen therapy,
* Hospitalization in the last 1 month,
* Patients with physical or mental health problems that would prevent communication were not included in the study.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Test- FVC | 0- 8. weeks
  Forced Vital Capacity (FVC): The amount of air that is exhaled forcefully and rapidly after taking as much breath as possible.
Respiratory Function Test- FEV1 | 0- 8. weeks
  1st Second Forced Expiratory Volume (FEV1): The amount of air exhaled in the first second of the FVC test.
Respiratory Function Test- FEF | 0- 8. weeks
  Forced Expiratory Flow (FEF): The average flow rate during the middle half of the FVC test.
Respiratory Function Test- PEFR | 0- 8. weeks
  Peak Expiratory Flow Rate (PEFR): The maximum airflow rate achieved during a forced exhalation.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankiri Karatekin University, Çankırı, Ori̇ji̇n, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No